CLINICAL TRIAL: NCT01645839
Title: Role of Intrathecal Chemotherapy With Liposomal Cytarabine (DepoCyte®) in Patients Wih Leptomeningeal Metastasis of Breast Cancer. A Randomized Phase III Study.
Brief Title: Interest of Intrathecal Chemotherapy With Liposomal Cytarabine (DepoCyte®) in Meningeal Metastasis of Breast Cancer
Acronym: DEPOSEIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEPOSEIN-1008; 2010-023134-23 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer; Leptomeningeal Metastases
Keywords: Leptomeningeal metastasis; Intrathecal chemotherapy; Depocyte
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic treatment with Depocyte (Experimental): Intrathecal injection of Liposomal Cytarabine (Depocyte®) every 14 ± 2 days for a total of 5 cycles and then every 28 ± 4 days until progression.
  Interventions: Drug: Liposomal Cytarabine
- Systemic treatment without Depocyte (No Intervention): No intrathecal injection.

INTERVENTIONS:
Drug: Liposomal Cytarabine — 50mg (5 mL) by slow intrathecal injection (1-5 minutes) directly into the cerebrospinal fluid (CSF) via a ventricular catheter directly into the lumbar sac during a lumbar puncture.
  Other Names: Depocyte; Aracytine
  Arms: Systemic treatment with Depocyte

SUMMARY:
The purpose of this study is to evaluate the impact of Depocyte® IT combined with the systemic standard treatment in terms of clinical and/or radiological neuromeningeal progression free survival (SSPN)

DETAILED DESCRIPTION:
After the signature of the consent form and validation of the eligibility inclusion criteria, patients will be randomized. Treatment will start within a maximum of 10 days after randomization.

Arm A: Systemic standard treatment without DepoCyte® Arm B: Systemic standard treatment with DepoCyte® DepoCyte® will be slowly administered by injection (1 to 5 minutes) of 50 mg (5 mL) into the CSF via a lumbar puncture or a ventricular device

* every 14 +/- 2 days for a total of 5 cycles (induction treatment)
* then every 28 +/-4 days until progression (maintenance treatment) Standard systemic treatment by chemotherapy, targeted therapy or hormonal therapy is at the discretion of the investigator taking into account the breast cancer sub-type and previous treatments. The systemic treatment will be determined before randomization. It can be modified at any time according to the treating oncologist. Focal radiotherapy to symptomatic sites is allowed. The usual follow-up of patients treated by IT DepoCyte® of every 14 days for the first two months and then monthly is not modified in patients of Arm B. Evaluation in Arm A will be matched to Arm B, and are thus more frequent than routinely done because such patients are usually seen every 3 weeks. The follow-up for systemic disease is left at the discretion of the treating oncologist.

Translational research Only Oscar Lambret Center will participate in this exploratory analysis. For patients who accept to participate, a 10 mL CSF sample will be collected at enrollment and once per month, just before treatment.

* Arm A: at monthly visit
* Arm B: at a IT injection, once per month, just before DepoCyte® injection Samples will be sent to the analysis center as soon as possible and will be destroyed at the end of all study-related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive breast cancer
* New diagnosis of leptomeningeal metastasis confirmed by CSF cytology, or by the combination of typical clinical symptoms or signs with typical MRI abnormalities
* Cerebrospinal MRI criteria: no visible lesion, or meningeal metastases <0.5 cm, or >0.5 cm largest diameter if focal radiotherapy planned
* Indication for systemic treatment (chemotherapy and/or targeted therapy and/or hormonal therapy) at the time of enrollment. Systemic treatment is at the discretion of the investigator (in collaboration with the treating oncologist if different) according to cancer characteristics, previous treatments, and clinical and biological disease characteristics. Focal radiotherapy is permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patients unable to walk due to a palsy but able to use a wheelchair are considered as ambulatory patients
* Expected survival of at least 2 months. Patients with rapidly progressive systemic disease are not eligible for this trial
* Co-existing asymptomatic brain metastases are permitted
* In case of suspicion of CSF flow block, or after focal radiotherapy for the treatment of a CSF flow block, a CSF flow study will be performed (isotopic method) to confirm the absence of CSF block
* Patients must have recovered from acute adverse events of other anticancer treatments previously administered
* Adequate bone marrow, renal, and hepatic function with the following range: bilirubin ≤ 3 x upper limit of normal (ULN), ASAT ≤ 2.5 x ULN or ≤ 5 x ULN in presence of liver metastases
* Adequate contraception (CPMP/ICH/286/95) for patients of reproductive potential (e.g., barrier method, vasectomy of partner, abstinence) (hormonal contraception not permitted)
* Patient affiliated to the French Social Security
* Able to understand the requirements of the study, date and sign written informed consent

Exclusion Criteria:

* Leptomeningeal metastasis related to other primary tumors than breast cancer
* History of other cancer (<5 years) except adequately treated cervical cancer, or basocellular or spinocellular skin cancer
* Contra-indication to MRI (including claustrophobia)
* MRI criteria: CSF flow obstruction (hydrocephalus on brain MRI or obstacle on spinal MRI)
* Contra-indication to lumbar puncture and to implantation of a ventricular device
* Progressive brain metastases thought to require whole brain radiotherapy
* Prior cranio-spinal irradiation (prior brain focal radiotherapy or whole brain radiotherapy for brain metastases permitted)
* Prior intrathecal chemotherapy or targeted therapy
* Prior systemic cytarabine treatment or prior systemic high-dose methotrexate treatment
* Concomitant systemic high-dose methotrexate treatment
* Ventriculo-peritoneal shunt
* Active infection (systemic or CNS)
* Hypersensitivity to cytarabine or DepoCyte
* Patient presenting with other severe non-controlled disease which could compromise the participation in the study (infection, cardio-vascular disease, gastro-intestinal disease, renal disease, pulmonary disease)
* Enrollment into another study evaluating a drug within 30 days before the screening visit
* Breast feeding woman or pregnancy. Nursing is not permitted for 6 months after the study
* Impossibility to adhere to the requirements of the study for geographic, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Leptomeningeal disease-related neurological progression-free survival (LM-PFS) | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  time between randomization and date of first leptomeningeal progression (defined according to clinical-neurological or imaging criteria) or date of death (death from any cause) whatever occurs first. Patients alive without neurological progression at the time of the last follow-up will be censored at the date of the last visit.

SECONDARY OUTCOMES:
Response of leptomeningeal metastases | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  Evaluated by clinical improvement, cytological improvement and MRI improvement. At 2 and 6 months, and best leptomeningeal disease response to treatment in response to treatment
Progression free survival (PFS) | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  PFS defined by the time between randomization and date of first progression: leptomeningeal, parenchymal, systemic (extra-CNS) or date of death (from any cause) if it occurs first. Patients alive and without progression at the time of the last follow-up will be censured at the date of the last visit. The different components of PFS will also be estimated considering the competing risk approach.
Overall survival | Until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  Time between the date of randomization in the study and the death of the patient (from any cause).
Tolerance to DepoCyte® according to NCI CTCAE V4.0 | Up to 30 days after the last administration of the study treatment
  Safety and tolerability profile of DepoCyte® according to NCI-CTCAE v4.0. Adverse events will be considered as severe if the grade is more than 2. All AE will be taken into account except events unequivocally related to the underlying disease or its progression. SAE will be also reported.
Q-TWiST | Calculated at the end of study
  Q-TWiSTanalysis defined by 3 health status: time with toxicity before progression (TOX), time after progression (PROG) considering progression at any site, and time without toxicity and without progression (TWiST).

OTHER OUTCOMES:
Quality of life (questionnaire QLQ C30, BN20 and C15) | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  Quality of life data will be described and compared between the 2 groups of treatment by estimating the impact of DepoCyte® in terms of time to definitive deterioration of quality of life will be also compared. A deterioration of quality of life is defined as by a decrease of 10 points of the quality of life score or an increase of 10 points for quality of life symptoms.
Autonomy in daily life (questionnaire Instrumental Activities in Daily Living) | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  IADL scale which evaluates the repercussions of the patients difficulties in the different activities of daily life.
Emotional state of the patient assessed by the psychological distress score | At baseline
  Emotional Distress Profile (EDP) scale and Patient Global Impression of Change (PGI-C) scale.
Identification and quantification of tumor cells in the CSF by the Veridex technique for the diagnosis and the follow-up of breast cancer leptomeningeal metastases | At baseline, then every 2 weeks for 2 months, after 2 months from baseline once a month until progression (up to 6 months) and at the end of the study (up to 6 months)
  60 samples analysed at the diagnostic and monitoring of tumor meningitis moments, by VERIDEX technique: the presence of tumours cells is affirmed if there is no more than 1 cell in 7.5 mL.
Leptomeningeal response according to RANO criteria combining clinical, CSF cytological and imaging response | Done at the end of study
  Leptomeningeal response according to RANO criteria combining clinical, CSF cytological and imaging response

CONTACTS AND LOCATIONS:
Overall Officials: Emilie LERHUN, MD, Principal Investigator — Centre Oscar Lambret
Locations (10):
- France (10):
  - Centre Hospitalier Universitaire Groupe Sud, Amiens
  - Centre Hospitalier Universitaire Lyon, Bron
  - Centre G.F. Leclerc, Dijon
  - CHU de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Antoine Lacassagne, Nice
  - Hôpital Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Rhun E, Wallet J, Mailliez A, Le Deley MC, Rodrigues I, Boulanger T, Lorgis V, Barriere J, Robin YM, Weller M, Bonneterre J. Intrathecal liposomal cytarabine plus systemic therapy versus systemic chemotherapy alone for newly diagnosed leptomeningeal metastasis from breast cancer. Neuro Oncol. 2020 Apr 15;22(4):524-538. doi: 10.1093/neuonc/noz201. PMID 31637444